CLINICAL TRIAL: NCT00825552
Title: Pharmacological Treatment of Children and Adolescents With Severe Mood Dysregulation. An Open Trial With Risperidone.
Brief Title: Pharmacological Treatment of Children and Adolescents With Severe Mood Dysregulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Luis Augusto Rohde, Federal University of Rio Grande do Sul, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 19091979
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Severe Mood Dysregulation
Keywords: Risperidone; Severe mood dysregulation; bipolar; children
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Risperidone — 0,5-4 mg/day for 8 weeks (twice a day)

SUMMARY:
The purpose of this study is to investigate whether Risperidone is effective in children and adolescents with severe mood dysregulation.

DETAILED DESCRIPTION:
Severe Mood Dysregulation(SMD) is a new construct in children and adolescents characterized by persistent and non episodic irritability, hyperarousal and emotional reactivity.

This is an open label trial using Risperidone in children and adolescents( 7-17 years old) diagnosed with SMD.

We hypothesized that Risperidone would improve externalizing symptoms as well as depressive and/or maniac symptomatology. We also consider the effect of the pharmacological intervention in the co-morbid disorders especially ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of Severe Mood Dysregulation
* 7-17 years
* IQ > 70

Exclusion Criteria:

* Bipolar disorder
* IQ<70
* Psychosis

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
We use as the primary outcome the subscale of irritability of the Aberrant Checklist Behavior which measures the intensity of irritability, temper tantruns and hyperarousal symptoms | 11/2010

CONTACTS AND LOCATIONS:
Overall Officials: Rohde A Luis, Phd, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Program of Bipolar Children and adolescents — http://www.ufrgs.br/procab